CLINICAL TRIAL: NCT07127419
Title: Effects of Music-Based Interventions on Sleep Patterns and Physiological Responses in Premature Newborns: A Systematic Review and Meta-Analysis
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sevgi Beyazgül, Sevgi Beyazgül, Istanbul University - Cerrahpasa
Other Study IDs: İstanbul Universty Cerrahpaşa
Record Dates: First submitted 2025-08-01; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Sleep; Newborn
Keywords: lullaby; music therapy; Sound-Based Interventions; newborn; sleep; preterm; term
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lullaby and/or Music Therapy Group: Other Sound-Based Interventions Group
- 1

SUMMARY:
Sleep in the neonatal period is a fundamental biological requirement for regulating growth, neurodevelopment, and the immune system. However, disruptions in sleep patterns during this period are common among both term and preterm infants. Preterm infants have a more fragile sleep structure due to incomplete neurological maturation, while term infants may also experience sleep difficulties during the postnatal adaptation process. Improving sleep onset and sleep quality in newborns is crucial for the well-being and quality of life of both the infant and the family.

DETAILED DESCRIPTION:
Music therapy-particularly lullabies-has been a traditional approach used for centuries to help infants fall asleep. It is believed that music and lullabies promote relaxation by regulating respiration and heart rate in infants, reducing stress responses, and thereby enhancing sleep quality. In recent years, there has been growing interest in music-based interventions in neonatal intensive care units, as these methods offer non-invasive, easily applicable, and cost-effective alternatives. However, research findings on the effects of music therapy and lullabies on neonatal sleep are varied. Due to the physiological and behavioral differences in preterm infants, their responses to music-based interventions may differ from those of term infants. Therefore, comprehensive evaluations of studies involving both preterm and term neonates are crucial for synthesizing current evidence and guiding healthcare professionals.

The aim of this systematic review and meta-analysis is to evaluate the effects of lullaby and music therapy interventions on sleep quality, sleep duration, and sleep onset latency in both preterm and term neonates, and to provide an up-to-date summary of the existing literature.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants who are clinically stable and between 26 and 37 weeks' gestational age.
* Infants monitored in the neonatal intensive care unit (NICU).
* A music-based intervention
* Sleep outcomes and/or physiological parameters measured.
* Randomised controlled design Full-text studies are available.

Exclusion Criteria:

* Non-neonatal infants (aged over 28 days). Term infants (≥37 weeks).

  * Non-neonatal age groups
  * Only assessing secondary outcomes, such as parental anxiety or caregiver stress
  * Case reports, conference abstracts, letters, etc.

Ages: 26 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This meta-analysis includes preterm (gestational age 26-37 weeks) neonates who were exposed to music therapy, lullabies, or other sound-based interventions in randomized controlled or quasi-experimental studies.
Sampling Method: Non-Probability Sample
Enrollment: 1415 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality in Neonates | During or within 24 hours after the intervention period
  - Weight gain Sleep-related indicators: sleep duration, duration of quiet sleep, sleep-wake cycle and brain activity, as measured by aEEG.